CLINICAL TRIAL: NCT00628277
Title: Methods of Weight Loss in Overweight Coronary Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator: Philip Ades MD, Professor of Medicine, University of Vermont college of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03-049
Record Dates: First submitted 2008-02-26; First posted 2008-03-05 (Estimated); Last update posted 2008-03-05 (Estimated); Status verified 2008-02

CONDITIONS: Obesity
Keywords: Obesity; coronary heart disease; coronary risk factors; weight loss; exercise
MeSH Terms: conditions — Obesity; Coronary Disease; Weight Loss; Motor Activity | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Arm 1: high caloric expenditure exercise plus dietary counseling
  Interventions: Behavioral: high caloric expenditure exercise
- 2 (Active Comparator): Arm 2: low caloric expenditure exercise plus dietary counseling
  Interventions: Behavioral: low caloric expenditure exercise plus dietary counseling

INTERVENTIONS:
Behavioral: high caloric expenditure exercise — high caloric expenditure exercise plus dietary counseling
  Arms: 1
Behavioral: low caloric expenditure exercise plus dietary counseling — low caloric expenditure exercise plus dietary counseling
  Arms: 2

SUMMARY:
We hypothesize that a combination of high-caloric expenditure exercise and behavioral weight loss counseling would lead to a greater loss of fat mass and a greater improvement in cardiometabolic risk factors that standard (lower caloric expenditure) cardiac rehabilitation exercise plus counseling.

DETAILED DESCRIPTION:
We hypothesize that a combination of high-caloric expenditure exercise and behavioral weight loss counseling would lead to a greater loss of fat mass and a greater improvement in cardiometabolic risk factors that standard (lower caloric expenditure) cardiac rehabilitation exercise plus counseling.

The study population consists of overweight (BMI >27) patients with established coronary heart disease. The exercise and counseling program was of 4 months duration with extended follow up at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Coronary heart disease
* BMI > 27
* Peak Vo2 > 14.4 ml/kg/min

Exclusion Criteria:

* Presence of diabetes

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2002-10; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Fat Mass | 4 months, 12 months

SECONDARY OUTCOMES:
Intrabdominal (visceral) fat | 4 months
Insulin stimulated glucose disposal | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Philip A Ades, MD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont College of Medicine, Burlington, Vermont, United States

REFERENCES:
- [Derived] Ades PA, Savage PD, Lischke S, Toth MJ, Harvey-Berino J, Bunn JY, Ludlow M, Schneider DJ. The effect of weight loss and exercise training on flow-mediated dilatation in coronary heart disease: a randomized trial. Chest. 2011 Dec;140(6):1420-1427. doi: 10.1378/chest.10-3289. Epub 2011 Jul 21. PMID 21778256
- [Derived] Ades PA, Savage PD, Toth MJ, Harvey-Berino J, Schneider DJ, Bunn JY, Audelin MC, Ludlow M. High-calorie-expenditure exercise: a new approach to cardiac rehabilitation for overweight coronary patients. Circulation. 2009 May 26;119(20):2671-8. doi: 10.1161/CIRCULATIONAHA.108.834184. Epub 2009 May 11. PMID 19433757